CLINICAL TRIAL: NCT06886763
Title: Assessment of Hepatocarcinoma Innervation by Tissue Transparisation and Pharmacological Screening
Brief Title: HCC Innervation Assessment
Status: Active, not recruiting | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL24_1190
Record Dates: First submitted 2025-03-14; First posted 2025-03-20 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Hepatocarcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | US Export: No

GROUPS / COHORTS (1):
- Patients with HCC candidates for hepatectomy or liver transplantation, with and without treatment
  Interventions: Other: Liver innervation markers

INTERVENTIONS:
Other: Liver innervation markers — Liver innervation markers will be quantified immediately after resection by transparisation technique.

SUMMARY:
Primary liver cancer casualties are ranked 3rd worldwide and are still on the rise despite the recent advent of adequate hepatitis B and C therapies. Genetic diseases of the liver and hepatic comorbidities, such as alcoholic liver disease and metabolic syndrome with metabolic-associated steatohepatitis, are long-term cooperators or independent factors fostering the onset of hepatocellular carcinoma (HCC) and enhancing disease heterogeneity. Though HCC is known to develop in 90% of cases of cirrhosis, its onset and clinical outcomes, in terms of phenotypes and speed of progression, are highly variable from one patient to another. Despite the identification of several potential therapeutic targets, most drugs have failed to exceed the efficacy of currently available compounds. Treatments with tyrosine kinase inhibitors for instance lead to short-term, unavoidable relapse, whereas treatment with immune checkpoints inhibitors or growth factors inhibitors currently provide some hope for only a minority of patients with unresectable HCC.

In this respect, cellular/tissular structures linking the general pathophysiology of the patient with HCC may be of interest, as they are patient-specific and may uncover novel ways of defining stratification criteria. In line with such notions, several recent original papers and related commentaries highlighted the relevance of studying cancer neurosciences of peripheral organs. In that context, pathological innervation and autonomous nervous system involvement or dysregulation have been identified in ovarian, prostate, gastric and pancreatic cancers, nurturing tumor stroma and conferring stronger carcinogenic properties. Moreover, the autonomic nervous system post-synaptic receptors have been shown to be favorably actionable in some experimental conditions in cancer.

The autonomic nervous system comprises the sympathetic (adrenergic signaling) and parasympathetic (cholinergic signaling) arms that relay signals both ways along the brain-liver neural axis in order to regulate involuntary functions of the body by adjusting its internal functions, after an external stimulus. The liver is an innervated organ that hosts autonomic afferent and efferent autonomic nervous system nerves, in constant communication with the central nervous system through the brainstem. Afferent and efferent nerves are made of adrenergic (relies on epinephrine or norepinephrine as its neurotransmitter, stress signal) and cholinergic (relies on acetylcholine as its neurotransmitter, resting signal) fibers that each convey mediators to regulate liver functions in real-time.

As a consequence, as also notably pointed out by Tracey's theory and evidence for cholinergic blockade of inflammation, these signals also regulate several processes that may directly or indirectly impact HCC onset and growth. However, data on the association between HCC and neural factors are scarce and sometimes conflicting. It was reported that portal hypertension, a recognized risk factor for HCC development and recurrence, is correlated with autonomic nervous system dysfunction. In addition, proliferation of hepatocytic progenitors, instrumental in HCC, is impaired by adrenergic signaling. Conversely, cholinergic signaling was shown to attenuate apoptosis in the mouse liver, and liver angiogenesis is under positive sympathetic regulation. Interestingly, human liver autonomic nervous system innervation is more developed than in rodents. Indeed, it extends deeper into the lobule, increasing its capacities of regulation. This latter notion suggests that autonomic nervous system-related mechanisms observed in animals may play more important roles in humans.

The primary goal of this study is to assess the innervation of tumor and peritumor tissues in HCC patients who undergo liver resection or liver transplant.

ELIGIBILITY:
Inclusion Criteria:

* Patients with hepatocarcinoma who undergo surgical resection or liver transplant
* Patients with and without treatment

Exclusion Criteria:

* - Pregnant or lactating women
* Minor patient
* Patient under legal protection measure or deprived of their liberty

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 300 patients with hepatocarcinoma who undergo surgical resection or liver transplant will be recruited at Hospitals of Lyon (GHN, GHS)
Sampling Method: Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2024-06-30 (Actual); Primary Completion 2029-04-30 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Assessment of morphological parameters (mature, immature, sympathetic and parasympathetic nerves) of innervation of peritumoral and tumor tissue using tissue transparisation (clearing) techniques. | Outcome measure will be assessed immediately after the surgery on fresh tissues. No follow-up is required.

CONTACTS AND LOCATIONS:
Locations (2):
- Groupement hospitalier Sud, Hospices Civils de Lyon, France, Egypt
- Groupement Hospitalier Nord, Hospices Civils de Lyon, France, France